CLINICAL TRIAL: NCT04834804
Title: Effects of a 12-week Suspension Versus Free Weight Training Program on Body Composition and Handgrip Strength in Older Men
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Bologna (Other)
Responsible Party: Principal Investigator, Francesco Campa, Principal investigator, University of Bologna
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 23032015
Record Dates: First submitted 2021-04-04; First posted 2021-04-08 (Actual); Last update posted 2021-04-09 (Actual); Status verified 2021-04

CONDITIONS: Effect of Different Exercise Programs on Body Composition
MeSH Terms: interventions — Exercise

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Suspension training group (Experimental)
  Interventions: Other: Physical activity
- Free weight training group (Experimental)
  Interventions: Other: Physical activity
- Control group (No Intervention)

INTERVENTIONS:
Other: Physical activity — 12 weeks of exercise training
  Arms: Free weight training group; Suspension training group

SUMMARY:
The present investigation lasted a total of 16 weeks, of which 4 were employed for assessment and measurements and 12 weeks were used for the exercise treatment. The participants underwent two different training programs carried out in three weekly 75-min sessions, on alternate days (Mondays, Wednesdays and Fridays, in the morning). Each session of both training programs consisted of a warm-up at the beginning and general stretching at the end. The exercises used in the suspension training program were: squat, rear deltoid row, biceps curl, chest press, low row, rotational ward, split squat whit Y deltoid fly, triceps pushdown. The exercises used in the free weight training program were: squat with support, unilateral squat, hip adduction and abduction, calves, hip flexor, alternating curl, French triceps press, and high row. Eleven participants were included in the control group.

ELIGIBILITY:
Inclusion Criteria:

* not having chronic disabling diseases
* not being bedridden institutionalized or hospitalized
* have their own mobility, without assistance from people, even if they have the aid of devices -without amputations.

Exclusion Criteria:

* the use of pacemakers and the presence of chronic and uncontrolled metabolic diseases

Min Age: 65 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 36 (Actual)
Dates: Start 2019-09-02 (Actual); Primary Completion 2019-12-02 (Actual); Study Completion 2019-12-02 (Actual)

PRIMARY OUTCOMES:
Body composition | 12 weeks
  Fat mass

CONTACTS AND LOCATIONS:
Locations (1):
- Francesco Campa, Bologna, Italy

IPD SHARING:
Plan to Share IPD: No